CLINICAL TRIAL: NCT02252640
Title: A Phase I/IIa Sporozoite Challenge Study to Assess the Safety and Protective Efficacy of Concomitant Administration of the Combination Malaria Vaccine Candidate Regimen of RTS,S/AS01¬B + ChAd63 and MVA Encoding ME-TRAP and Also RTS,S/AS01B Alone
Brief Title: A Safety and Efficacy Study of Concomitant Administration of ChAd63/MVA ME-TRAP + RTS,S
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC059; 2014-001301-40 (EudraCT Number)
Record Dates: First submitted 2014-09-25; First posted 2014-09-30 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Plasmodium Falciparum; Malaria; Vaccine; Plasmodium; Falciparum
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 (Active Comparator): Week 0: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01), Week 4: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01), Week 8: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01), Week 11: Controlled Human Malaria Infection (CHMI), Week 31-39: Repeat CHMI of sterilely protected volunteers.
  Interventions: Biological: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01)
- Group 2 (Active Comparator): Week 0: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01), Week 4: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01), Week 8: RTS,S/AS01B (10mcg of RTS,S and 1/5 of the standard dose of AS01), Week 11: Controlled Human Malaria Infection (CHMI), Week 31-39: Repeat CHMI of sterilely protected volunteers.
  Interventions: Biological: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01); Biological: RTS,S/AS01B (10mcg of RTS,S and one fifth of the standard dose of AS01)
- Group 3 (Active Comparator): Week 0: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01) & ChAd63 ME-TRAP (5 x 10^10 vp), Week 4: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01) & MVA ME-TRAP (2 x 10^8 pfu), Week 8: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01) & MVA ME-TRAP (2 x 10^8 pfu), Week 11: Controlled Human Malaria Infection (CHMI), Week 31-39: Repeat CHMI of sterilely protected volunteers.
  Interventions: Biological: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01); Biological: ChAd63 ME-TRAP (5 x 10^10 vp); Biological: MVA ME-TRAP (2 x 10^8 pfu)
- Group 4 (Active Comparator): Week 0: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01) & ChAd63 ME-TRAP (5 x 10^10 vp), Week 4: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01) & MVA ME-TRAP (2 x 10^8 pfu), Week 8: RTS,S/AS01B (10mcg of RTS,S and 1/5 of the standard dose of AS01) & MVA ME-TRAP (2 x 10^8 pfu), Week 11: Controlled Human Malaria Infection (CHMI), Week 31-39: Repeat CHMI of sterilely protected volunteers.
  Interventions: Biological: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01); Biological: RTS,S/AS01B (10mcg of RTS,S and one fifth of the standard dose of AS01); Biological: ChAd63 ME-TRAP (5 x 10^10 vp); Biological: MVA ME-TRAP (2 x 10^8 pfu)
- Group 5 (No Intervention): Week 11: Controlled Human Malaria Infection
- Group 6 (No Intervention): Week 31-39: Controlled Human Malaria Infection

INTERVENTIONS:
Biological: RTS,S/AS01B (50mcg of RTS,S and standard adult dose of AS01)
  Arms: Group 1; Group 2; Group 3; Group 4
Biological: RTS,S/AS01B (10mcg of RTS,S and one fifth of the standard dose of AS01)
  Arms: Group 2; Group 4
Biological: ChAd63 ME-TRAP (5 x 10^10 vp)
  Arms: Group 3; Group 4
Biological: MVA ME-TRAP (2 x 10^8 pfu)
  Arms: Group 3; Group 4

SUMMARY:
The purpose of this study is to assess two types of new malaria vaccines in different combinations. The study will enable us to assess:

1. The ability of the vaccines to prevent malaria infection.
2. The safety of the vaccines in healthy participants.
3. The response of the human immune system to the vaccines.

We will do this by giving 48 participants three sets of vaccinations over 8 weeks, then exposing them to malaria infection by allowing mosquitoes infected with malaria to bite under carefully regulated conditions. We will follow participants closely to observe if and when they develop malaria. If the vaccine combination provides some protection against malaria, participants will take longer to develop malaria than usual or will not develop malaria at all. We will also recruit 4 individuals to be control subjects - these participants won't receive any vaccinations but will be challenged with malaria.

Vaccinated volunteers who do not develop malaria infection in the blood after being infected with malaria by mosquito bite the first time may be invited back to be again infected with malaria in a repeat challenge experiment. This would happen approximately 5-7 months after the first challenge. The purpose of this second challenge will be to see how long the protection of the investigational vaccine against malaria lasts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner.
* Women only: Must practice continuous effective contraception for the duration of the study.
* Agreement to refrain from blood donation during the course of the study and for at least 3 years after the end of their involvement in the study.
* Written informed consent to participate in the trial.
* Reachable (24/7) by mobile phone during the period between Controlled Human Malaria Infection (CHMI) and completion of antimalarial treatment.
* Willingness to take a curative anti-malaria regimen following CHMI.
* For volunteers not living in Oxford: agreement to stay in a hotel room close to the trial centre during a part of the study (from at least day 6.5 post mosquito bite until anti-malarial treatment is completed).
* Answer all questions on the informed consent quiz correctly.

Exclusion Criteria:

* History of clinical malaria (any species).
* Travel to a malaria endemic region during the study period or within the preceding six months with significant risk of malaria exposure.
* Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin)
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data. If any volunteers in Group 1-4 undergo rechallenge, this exclusion criterion does not extend to the vaccines previously received in this trial
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (e.g. egg products, Kathon) or malaria infection.
* Any history of anaphylaxis post vaccination.
* History of clinically significant contact dermatitis.
* History of sickle cell anaemia, sickle cell trait, thalassaemia or thalassaemia trait or any haematological condition that could affect susceptibility to malaria infection.
* Pregnancy, lactation or intention to become pregnant during the study.
* Use of medications known to cause prolongation of the QT interval and existing contraindication to the use of Malarone
* Use of medications known to have a potentially clinically significant interaction with Riamet and Malarone
* Any clinical condition known to prolong the QT interval
* History of cardiac arrhythmia, including clinically relevant bradycardia
* Disturbances of electrolyte balance, eg, hypokalaemia or hypomagnesaemia
* Family history of congenital QT prolongation or sudden death
* Contraindications to the use of all three proposed anti-malarial medications; Riamet, Malarone and Chloroquine.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 standard UK units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
* An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system.59
* Positive family history in 1st and 2nd degree relatives <50 years old for cardiac disease.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of a combination immunization regimen with ChAd63/MVA ME-TRAP given concomitantly with RTS,S/AS01B against malaria sporozoite challenge. | 6 months
  Use statistical analysis to compare number of completely protected individuals (those who do not, by Day 23 following sporozoite challenge, develop blood stage infection measured by occurrence of P. falciparum parasitemia, assessed by blood slide)
Safety of a combination immunization regimen with ChAd63/MVA ME-TRAP given concomitantly with RTS,S/AS01B against malaria sporozoite challenge. | 6 months
  Occurrence of solicited and unsolicited adverse events will be monitored. Solicited and unsolicited AE data will be collected at each clinic visit. It will be collected from diary cards, clinical review, clinical examination (including observations) and laboratory results. This AE data will be tabulated and frequency, duration and severity of AEs compared between groups.

SECONDARY OUTCOMES:
Immunogenicity generated in malaria naïve individuals of two different dosing regimens of RTS,S/AS01B given concomitantly with ChAd63/MVA ME-TRAP, and of RTS,S/AS01B alone at either full standard dose or with a reduced third dose. | 6 months
  To document immunogenicity measures, capturing humoral and cellular immune responses to both ChAd63/MVA ME-TRAP and RTS,S as follows: Anti-CS (RT, C-term, full-length), anti-HBs, and anti-ME-TRAP antibody titers; frequency of CS-specific, HBs-specific, and TRAP and ME specific T cells; ChAd63 neutralizing antibody titers; avidity index of anti-CS antibodies. To undertake exploratory analysis of the correlation of these measures with vaccine efficacy. To, furthermore, undertake an exploratory analysis of transcriptomic correlates of vaccine immunogenicity and efficacy. This may be undertaken by microarray analysis or RNA sequencing or both techniques.

OTHER OUTCOMES:
Long term protective efficacy of a combination immunization regimen with ChAd63/MVA ME-TRAP given concomitantly with RTS,S/AS01B | 12 months
  Long term efficacy of the Group 1, 2, 3 and 4 vaccination regimens will be assessed by re-challenging any sterilely protected individuals at 5 - 7 months after the first CHMI and comparing the number of re-challengees who develop blood stage infection, and the time between CHMI and blood stage infection, with unvaccinated controls.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, Principal Investigator — University of Oxford
Locations (4):
- United Kingdom (4):
  - NIHR WTCRF, University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford, Oxfordshire
  - Surrey Clinical Research Centre, University of Surrey, Guildford, Surrey
  - NIHR/Wellcome Trust Imperial CRF, Hammersmith Hospital, Imperial College NHS Trust, London